CLINICAL TRIAL: NCT00790478
Title: Melatonin and Ulcerative Colitis: A Pilot Clinical Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Paul D Terry PhD, Principal Investigator, Emory University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00008173; IBD-0223
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Melatonin; Gastrointestinal; Irritable Bowel syndrome; Sleep; Pilot Study
MeSH Terms: conditions — Colitis, Ulcerative; Irritable Bowel Syndrome | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo -- lactose pill.
  Interventions: Other: Placebo
- Melatonin (Active Comparator): Melatonin
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Study Pill (5 mg/d) taken once daily, preferably an hour before bedtime, for 12 weeks.
  Arms: Melatonin
Other: Placebo — Study Placebo taken once daily, preferably an hour before bedtime, for 12 weeks.
  Arms: Placebo

SUMMARY:
Ulcerative colitis is an inflammatory bowel disease that afflicts up to one million people in the U.S. Symptoms include rectal urgency, bloody diarrhea, moderate to severe abdominal pain, fever, and fatigue. Melatonin is a hormone that is associated with sleep and other body functions that may be related to health. Melatonin is produced in the pineal gland and, in fact, it is produced in even greater amounts in the gut. Melatonin appears to be important in gastrointestinal tract physiology and health, and data from cell and animal experiments, and some studies in humans, suggest that supplemental melatonin may help ameliorate colitis. Given that current treatments for ulcerative colitis are not always effective, and often have serious side effects, there is considerable interest in finding alternative treatments for this disease. However, experimental data on the ability of melatonin to improve ulcerative colitis in humans are lacking. To address this, we plan to conduct a pilot clinical trial (60 adult male and female participants) that will obtain preliminary data about the effectiveness of melatonin supplementation as a treatment for ulcerative colitis in adult men and women with the disease.

The "Melatonin and Ulcerative Colitis" study funded by a grant from the Broad Foundation's Broad Medical Research Program (http://www.broadmedical.org).

DETAILED DESCRIPTION:
Problem of Interest:

Current treatments for ulcerative colitis are not always effective, and often have serious side effects. Therefore, there is considerable interest in finding alternative treatments for this disease. Physiologic data suggest that melatonin is important in gastrointestinal (GI) tract physiology and health, and data from in vitro studies, animal experiments, and some studies in humans suggest that supplemental melatonin may have an ameliorative effect on colitis. However, experimental data on the ability of melatonin to improve ulcerative colitis in humans are lacking. The long-term goal of this proposal is to examine whether melatonin supplementation helps alleviate mild-to-moderate colitis symptoms. To this end, we plan to conduct a pilot randomized, double-blind, placebo-controlled trial (n = 60) that will obtain preliminary data about the effectiveness of melatonin supplementation as a treatment for ulcerative colitis in adult men and women with mild to moderate flare-up of the disease. The specific aims of the trial are: (i) to estimate the effect of 12 weeks of 5 mg/day supplementation with melatonin on ulcerative colitis remission, (ii) to estimate the effects of melatonin supplementation on tissue levels of cytokines and other markers of inflammation, (iii) to determine whether melatonin's effects vary according to baseline (endogenous) melatonin levels, (iv) to determine the feasibility of recruiting and retaining a sufficient number of ulcerative colitis patients for a larger, more definitive study, and (v) to determine whether melatonin supplementation has any adverse side-effects when taken daily for 12 weeks in adults with ulcerative colitis.

How the Problem Will Be Studied:

The overall study design of this trial is that of a randomized, double-blind, placebo-controlled clinical trial. Patients will be recruited from those seeing their IBD clinicians at one of three study sites: Emory University, Atlanta Gastroenterology Associates, or the Atlanta VA Medical Center. Eligibility will be based first on the severity of disease, determined by physician exam, and through sigmoidoscopy (as part of the Mayo Scoring System). The Project Coordinator will meet with patients to further determine eligibility, as there are restrictions based on age, medical history, medications taken, pregnancy, and others. Willing patients who are otherwise eligible at that point will undergo a one-week placebo run-in to assess compliance and any reported side-effects. Eligible patients will undergo their first study sigmoidoscopy, will provide biological samples for processing (blood, urine, and rectal biopsy tissue), and will be randomized into treatment (5 mg/d at bedtime) or placebo (also at bedtime). They will be given sleep logs and symptoms logs to fill out weekly during the trial, and they will fill out a colitis-related quality of life questionnaire. They will be called once per week by the Project Coordinator to check on the study participants, to assess compliance and side-effects, and to answer any questions. There will be a clinical visit two weeks after randomization, to assess symptoms and any side effects. The next scheduled clinical visit is at the end of the trial, where another sigmoidoscopy and sample collection will take place. Any other interim clinical visit will be at the discretion of the patients and his or her study physician. Lastly, patients will complete a questionnaire about colitis-related quality of life during the trial and will be asked as to whether they suspected which treatment arm they were in. The following period will be devoted to data analysis, publication of study results, and closeout. Please see attached protocol for details.

Importance of the Knowledge to be Gained:

The proposed research will have both public health and scientific importance. Ulcerative colitis is not a rare condition, and sufferers often deal with debilitating symptoms. Thus, a greater understanding of ways of treat ulcerative colitis would be of potential relevance to a great number of people.

How the Research Will Advance Scientific Knowledge and/or Human Health

UC is a common gastrointestinal disorder in adults, one that can have debilitating symptoms and severe health consequences. Current treatments are not always effective, and often have serious side effects. Therefore, there is considerable interest in finding alternative treatments for this disease. Physiologic data suggest that melatonin is important in GI tract physiology and health, and data from in vitro studies, animal experiments, and some studies in humans, suggest that supplemental melatonin may have an ameliorative effect on colitis. Given our newly-funded pilot clinical trial was awarded the maximum funding available from the Broad Foundation, with no funds allocated to explore potentially important biological mechanisms, we feel that this is an excellent opportunity to validate potential clinical benefits of melatonin as an adjunctive therapy for UC in humans, with mechanistic insights into the various levels of the inflammatory process that may be influenced by melatonin in vivo. Thus, the proposed study is a) innovative, b) supported by experimental data, and c) may ultimately lead to improved treatment of UC based on clinical and mechanistic knowledge gained through this study conducted in human patients.

To date, there has been no formal clinical trial of melatonin therapy for UC in humans, and there have been few mechanistic investigations into the potential mode of action of this compound on the pathomechanisms identified thus far. Given the very low toxicity documented for even high levels of melatonin in animals and human subjects, this relatively inexpensive treatment may represent an attractive alternative for patient suffering from mild to mid-grade UC given the low incidence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years.
* Diagnosed with ulcerative colitis and currently experiencing a flare up of mild-moderate severity according to Mayo Scoring system (>=4 and <=10).
* Has a regular GI physician(s).
* Availability for 14 weeks after enrolling in the study.
* Female patients of child bearing potential must be surgically sterile or have a negative urine pregnancy test and practice acceptable contraception (i.e., abstinence, oral, intramuscular, or implanted hormonal contraception, 2-barrier methods such as condom, diaphragm or spermicide).

Exclusion Criteria:

* Night shift workers; otherwise, inability to attend morning study visits.
* Current severe colitis according to the Mayo Scoring System (>10) or requiring hospital admission, or current very mild colitis (<4).
* Current supplemental intake of melatonin or currently using tobacco products.
* Proctitis or Crohn's disease
* Previous gastrectomy or small or large bowel resection
* Malabsorption syndrome (e.g., pancreatic insufficiency).
* History of large bowel resection for any reason.
* Diagnosed narcotic or alcohol dependence.
* On renal dialysis.
* Active liver disease (a chronic condition or under current therapy)
* Seizure disorders
* Immune system disorders
* Any history of hypo- or hyperparathyroidism.
* Unable to be off aspirin for 7 days.
* Use of systemic or rectal steroids in the past 8 weeks.
* Have a history of allergy or hypersensitivity to melatonin.
* History of bleeding disorder or current use of anticoagulant medication.
* Current use of calcium channel blockers, anticonvulsants, sedatives, hypnotics, or psychotropic medications.
* Women who are pregnant, breast-feeding, attempting conception, or planning to attempt conception over the following 6 months, or are currently taking hormone replacement therapy (HRT).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Consultative Gastroenterology, Atlanta, Georgia

REFERENCES:
- [Background] D'Haens G, Sandborn WJ, Feagan BG, Geboes K, Hanauer SB, Irvine EJ, Lemann M, Marteau P, Rutgeerts P, Scholmerich J, Sutherland LR. A review of activity indices and efficacy end points for clinical trials of medical therapy in adults with ulcerative colitis. Gastroenterology. 2007 Feb;132(2):763-86. doi: 10.1053/j.gastro.2006.12.038. Epub 2006 Dec 20. No abstract available. PMID 17258735
- [Background] von Gall C, Stehle JH, Weaver DR. Mammalian melatonin receptors: molecular biology and signal transduction. Cell Tissue Res. 2002 Jul;309(1):151-62. doi: 10.1007/s00441-002-0581-4. Epub 2002 May 18. PMID 12111545
- [Background] Li JH, Yu JP, Yu HG, Xu XM, Yu LL, Liu J, Luo HS. Melatonin reduces inflammatory injury through inhibiting NF-kappaB activation in rats with colitis. Mediators Inflamm. 2005 Aug 31;2005(4):185-93. doi: 10.1155/MI.2005.185. PMID 16192667
- [Background] Nosal'ova V, Zeman M, Cerna S, Navarova J, Zakalova M. Protective effect of melatonin in acetic acid induced colitis in rats. J Pineal Res. 2007 Apr;42(4):364-70. doi: 10.1111/j.1600-079X.2007.00428.x. PMID 17439553
- [Background] Song GH, Leng PH, Gwee KA, Moochhala SM, Ho KY. Melatonin improves abdominal pain in irritable bowel syndrome patients who have sleep disturbances: a randomised, double blind, placebo controlled study. Gut. 2005 Oct;54(10):1402-7. doi: 10.1136/gut.2004.062034. Epub 2005 May 24. PMID 15914575
- [Background] Maldonado MD, Calvo JR. Melatonin usage in ulcerative colitis: a case report. J Pineal Res. 2008 Oct;45(3):339-40. doi: 10.1111/j.1600-079X.2008.00584.x. Epub 2008 Mar 10. No abstract available. PMID 18331546
- [Background] Lu WZ, Gwee KA, Moochhalla S, Ho KY. Melatonin improves bowel symptoms in female patients with irritable bowel syndrome: a double-blind placebo-controlled study. Aliment Pharmacol Ther. 2005 Nov 15;22(10):927-34. doi: 10.1111/j.1365-2036.2005.02673.x. PMID 16268966
- [Background] Saha L, Malhotra S, Rana S, Bhasin D, Pandhi P. A preliminary study of melatonin in irritable bowel syndrome. J Clin Gastroenterol. 2007 Jan;41(1):29-32. doi: 10.1097/MCG.0b013e31802df84c. PMID 17198061

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated. No data were analyzed and data have since been destroyed.
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated. No data were analyzed, and data have since been destroyed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Melatonin | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Estimate Treatment Effect of 12 Weeks of 5 mg/Day Supplementation With Melatonin on UC Remission, and to Use the Estimate of This Effect and Its Variability to Calculate the Sample Size Needed for a Presumably Larger and More Definitive Trial.
Time Frame: April 2010
Population: Study was terminated. No data were analyzed, and data have since been destroyed.
Groups:
- Placebo: Placebo
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Investigate Whether Responses to Treatment Vary According to Certain Other Factors, Such as Age, Sex, Duration of Disease, Clinical Symptoms, Sleep Duration and Quality During the Trial, and Baseline Endogenous Melatonin.
Description: Study was terminated. No data were analyzed, and data have since been destroyed.
Time Frame: April 2010
Population: Study was terminated. No data were analyzed, and data have since been destroyed.
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Study was terminated. No data were analyzed, and data have since been destroyed.
Arm/Group | Melatonin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No